CLINICAL TRIAL: NCT02020681
Title: Effect of Curodont Repair or Placebo on the Remineralisation in Patients With Class 5 Carious Lesions: A Mono-centre, Split-mouth, Double-blinded, Placebo Controlled, Randomised, Post Marketing Clinical Study
Brief Title: Effect of Curodont Repair or Placebo on the Remineralisation in Patients With Class 5 Carious Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Credentis AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P11-4-CURAF; 14934.1 PFLS-LS (Other Grant/Funding Number: Swiss Committee for Technology and Innovation KTI)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Dental Caries
Keywords: Dental caries; Curodont Repair; P11-4
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curodont Repair (Experimental): Single application of Curodont Repair on treatment day D0 followed by a single application of fluoride (Duraphat) on D90.
  Interventions: Device: Curodont Repair; Device: Fluoride
- Placebo (Placebo Comparator): Single application of Placebo on treatment day D0 followed by a single application of fluoride (Duraphat) on D90.
  Interventions: Other: Placebo; Device: Fluoride

INTERVENTIONS:
Device: Curodont Repair — Self-assembling peptide, biomimetic re-mineralisation
  Other Names: P11-4
  Arms: Curodont Repair
Other: Placebo — Formulation of Curodont Repair without the peptide P11-4
  Arms: Placebo
Device: Fluoride — Single application on day D90

SUMMARY:
The purpose of this study is to evaluate the therapeutic benefit of Curodont Repair for the treatment of early buccal carious lesions compared to placebo.

DETAILED DESCRIPTION:
All study participants must have two early class V carious lesions in need of a treatment but not of an invasive treatment (split-mouth design). One lesion will be treated with Curodont Repair and one with placebo as control (single application). 3 months later fluoride (Duraphat) will be applied on both lesions. Study duration is 9 months. For assessment visual and tactile evaluation, pictures, ECM, Diagnodent Pen, Canary System, VAS is used.

ELIGIBILITY:
Inclusion Criteria:

* Two class V carious lesions which do not require an invasive treatment
* Size and form of the lesions: the lesions must both be fully visible and assessable and accessible
* Patients must be able and willing to observe good oral hygiene throughout the study

  -≥ 20 teeth
* Permanent dentition and ≤ 65 years
* Willing and able to attend the on-study visits
* Willing and able to understand all study-related procedures
* Written informed consent before participation in the study
* Negative pregnancy test for women of childbearing potential

Exclusion Criteria:

* The two study lesions must not be on adjacent teeth
* No adjacent restoration on study tooth surface
* Fluoride varnish application < 6 months prior to study treatment
* Patient suffers from diabetes
* Evidence of tooth erosion (due to excessive acidic drink consumption or reflux)
* History of head and neck illnesses (e.g. head/neck cancer)
* Any pathology or concomitant medication affecting salivary flow or dry mouth
* Any metabolic disorders affecting bone turnover
* Concurrent participation in another clinical trial with an investigational drug or device or participation in another clinical trial with an investigational drug or device within 30 days prior to study entry
* Pregnant and lactating woman

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is the difference of the change in the lesion size assessed by morphometry (standardised pictures) between investigational medical device and placebo group. | D0, D30, D90, D270
  Change of lesion size relative to baseline between study groups and different time points

SECONDARY OUTCOMES:
Difference in the change of Diagnodent Pen values between investigational medical device and placebo group. | D0, D30, D90, D180, D270
  only descriptively analysed
Change in lesion's progression assessed by VAS between investigational medical device and placebo group. | D0, D30, D90, D180, D270
  only descriptively analysed

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Krejci, Prof. Dr., Principal Investigator — University of Geneva
Locations (1):
- University of Geneva - Devision of Cariology and Endodontology, Geneva, Switzerland